CLINICAL TRIAL: NCT01782196
Title: A Phase II Multi Centre Study to Assess the Safety and Performance of Two Prototype One Piece Pouches in Subjects With an Ileostomy
Acronym: U366
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Leakage
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CC-0512-12-U366
Record Dates: First submitted 2012-12-19; First posted 2013-02-01 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Ileostomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Type A Pouch followed by Type B pouch (Experimental): Enhanced one piece drainable pouch with Type A mouldable adhesive for Stage 1 and 2 followed by pouch with Type B mouldable adhesive for Stage 3
  Interventions: Device: Enhanced one piece drainable pouch with Type A mouldable adhesive; Device: Enhanced one piece drainable pouch with Type B mouldable adhesive
- Type B Pouch followed by Type A pouch (Experimental): Enhanced one piece drainable pouch with Type B mouldable adhesive for Stage 1 and 2 followed by pouch with Type A mouldable adhesive for Stage 3
  Interventions: Device: Enhanced one piece drainable pouch with Type A mouldable adhesive; Device: Enhanced one piece drainable pouch with Type B mouldable adhesive

INTERVENTIONS:
Device: Enhanced one piece drainable pouch with Type A mouldable adhesive
Device: Enhanced one piece drainable pouch with Type B mouldable adhesive

SUMMARY:
Certain research and innovation projects require an assessment of the adhesive properties of adhesives, which cannot be established from in-vitro testing. The most valuable data for assessments of this type comes from adhesion and wear time studies involving application to living human skin on volunteers. The purpose of the study is to assess the safety and performance of an enhanced one piece drainable pouch with a mouldable skin barrier wafer in a group of subjects with an ileostomy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who provide written informed consent.
* Subjects who have an ileostomy and be over 18 years of age.
* Subjects who are currently using a one piece drainable pouch.
* Subjects who have unbroken peri-stomal skin (healthy normal skin defined as "normal unbroken skin with certain variations normal for this subject" to L1 on the SACs Instrument Scale).
* Subjects with a stoma considered 'normal' in appearance in accordance with the stoma, colour, moisture and structure rating scales.
* Subjects who are willing to attend clinic for a maximum of 5 separate occasions for scheduled visits.
* Subjects who are willing to discontinue the use of pastes, adhesive strips and rings/seals used to seal the area between the skin barrier wafer and stoma during the use of the study device.
* Subjects who other than their ileostomy considered to have a healthy/stable health status.
* Subjects who have good manual dexterity and be able to take care of their stoma independently, or have a consistent care provider.
* Subjects who are willing and able to complete a diary card for the duration of the study.

Exclusion Criteria:

* Subjects with a history of sensitivity to any one of the ostomy products or the components being studied.
* Subjects with stoma duration of less than 3 months.
* Subjects who currently use a belt with their usual appliance.
* Subjects who have been entered into the study before, or who have previously taken part in a study in the last month.
* Subjects who require convexity or other skin fillers (pastes, rings, seals) to even undulations of the skin.
* Subjects undergoing chemotherapy or radiotherapy.
* Subjects who have any other medical condition which, according to the investigator justifies exclusion from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety - evaluated by the nature and frequency of adverse events including stomal and peristomal skin condition and lesions | 59 days
  The primary objective of this study is to evaluate the safety of the enhanced one piece drainable pouch with a mouldable skin barrier wafer and two alternate adhesives in subjects with an ileostomy.

SECONDARY OUTCOMES:
Performance | 59 days
  Performance will be evaluated by comparing the following categories to the subject's usual pouching system
  Wear time Adhesion Ease of Use Mouldability Comfort and flexibility Security Skin protection Wafer seal integrity Undermining Filter performance Accessory usage
  At the end of the study a comparative assessment of the subject's usual pouching system and the study pouch will be made.

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Princess of Wales Hospital, Bridgend, Mid Glam
  - Wrexham Maelor Hospital, Wrexham, North Wales
  - Musgrove Park Hospital, Taunton, Somerset
  - Manor Hospital, Walsall, West Midlands
  - Homerton University Hospital, London